CLINICAL TRIAL: NCT03518177
Title: Comparison of the Effectiveness of Home and Supervised Pulmonary Rehabilitation in Candidate Patients With Bronchoscopic Lung Volume Reduction
Brief Title: Comparison of the Effectiveness of Home and Hospital-based PR in Candidate Patients With BLVR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, esra pehlivan, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: esra pehlivan
Record Dates: First submitted 2018-04-25; First posted 2018-05-08 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Emphysema; Bronchoscopic Lung Volume Reduction; Hospital-based Pulmonary Rehabilitation; Home-based Pulmonary Rehabilitation
MeSH Terms: conditions — Emphysema

STUDY DESIGN:
Intervention Model Description: Two parallel groups will be formed from patients with hospital-based pulmonary rehabilitation (Group 1) and those with home-based pulmonary rehabilitation(Group 2).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hospital-based PR group (Experimental): The patient will receive an 8-week supervised Pulmonary Rehabilitation Exercise Program at hospital
  Interventions: Other: Hospital-based pulmonary rehabilitation
- Home-based PR group (Experimental): The patient will receive an 8-week Pulmonary Rehabilitation Exercise Program at home
  Interventions: Other: Home-based pulmonary rehabilitation

INTERVENTIONS:
Other: Hospital-based pulmonary rehabilitation — The patient will receive an 8-week Pulmonary Rehabilitation Exercise Program including breathing exercises, treadmill walking, cycle ergometer, arm ergometer training and strengthening trainning with free weights at hospital.
  Arms: Hospital-based PR group
Other: Home-based pulmonary rehabilitation — The patient will receive an 8-week Pulmonary Rehabilitation Exercise Program including breathing exercises, free-walking, and strengthening training with free weights at home
  Arms: Home-based PR group

SUMMARY:
The recent years, the use of bronchoscopic lung volume reduction in emphysema patients instead of surgical operations has become widespread. Before this procedure, the implementation of Pulmonary Rehabilitation became a necessity. The inadequacy of the number of Pulmonary Rehabilitation Centers in our country and in our city and the increasing number of mentioned operations have increased the need for different exercise program applications. Prior to valve and coil applications in our study, changes in clinical conditions of patients will be examined if Pulmonary Rehabilitation is performed at home or in a hospital.

DETAILED DESCRIPTION:
The records of emphysema patients referred to the Pulmonary Rehabilitation Unit for prophylactic pulmonary rehabilitation prior to bronchoscopic lung volume reduction will be recorded prospectively. Two parallel groups will be formed from patients with hospital-based pulmonary rehabilitation (Group 1) and those with home-based pulmonary rehabilitation (Group 2). The patient will receive an 8-week Pulmonary Rehabilitation Exercise Program and will be reevaluated after 8 weeks. The differences in the parameters of initial and rehabilitation end-tracing and the differences between the groups will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Patients with emphysema and bronchoscopic lung volume reduction procedures decided by chest physician
* Acceptance of participation in a 2-month Pulmonary Rehabilitation program.

Exclusion Criteria:

-Possible orthopedic, cardiovascular or psychological disturbance that may prevent exercising.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline distance covered in six-minute walk test at 8 weeks | 8 weeks
Change from baseline modified Medical Council Dyspnea score at 8 weeks | 8 weeks
  The scale will rate the sensation of dyspnea as the person perceives it.The severity of dyspnea is rated on a scale of 0 to 4."0 point" means no dyspnea perception and "4point" means severe dyspnea perception.
Change from baseline Chronic Obstructive Airway Disease assesment test(CAT) score at 8 weeks | 8 weeks
  The COPD Assessment Test (CAT) is a questionnaire for people with COPD. It is designed to measure the impact of COPD on a person's life, and how this changes over time. Range of CAT scores from 0-40. Higher scores denote a more severe impact of COPD on a patient's life.
Change from baseline Forced Expiratory Volume in 1 second (FEV1) at 8 weeks | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Yedikule Chest Disease Hospital, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pehlivan E, Yazar E, Balci A, Turan D, Demirkol B, Cetinkaya E. A comparative study of the effectiveness of hospital-based versus home-based pulmonary rehabilitation in candidates for bronchoscopic lung volume reduction. Heart Lung. 2020 Nov-Dec;49(6):959-964. doi: 10.1016/j.hrtlng.2020.06.011. Epub 2020 Jul 21. PMID 32709500